CLINICAL TRIAL: NCT05391620
Title: Acute Effects of the 3/7 Method and 3X9 Method in Resistance Training on Testosterone, Glucocorticoid Cortisol, Growth Hormone and Lactate in Heart Failure and Coronary Artery Disease During Cardiac Rehabilitation
Brief Title: The Effect of the 3/7 vs 3X9 Method in Resistance Training on Metabolic Stress in Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Alexis Gillet, Principal Investigator, Université Libre de Bruxelles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2020276
Record Dates: First submitted 2022-04-07; First posted 2022-05-26 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure; Resistance Training; Coronary Artery Disease
Keywords: Cardiac rehabilition; exercise therapy; metabolic stress
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD group (Experimental): Coronary artery diseases
  Interventions: Other: Cardiac rehabilitation with 3/7 method; Other: Cardiac rehabilitation with 3X9 method
- HFrEF group (Experimental): Heart Failure with reduced Ejection Fraction
  Interventions: Other: Cardiac rehabilitation with 3/7 method; Other: Cardiac rehabilitation with 3X9 method

INTERVENTIONS:
Other: Cardiac rehabilitation with 3/7 method — HIIT ( 2 min 80% wmax: 2 min 50% wmax) during 30 minutes 3/7 method 3 rep (15 sec of rest), 4 rep (15 sec), 5 rep (15 sec), 6 rep (15 sec), 7 rep. (total volume : 25 repetitions) at 70 of 1 repetition Leg press, Dips Press, Leg curl, Traction and Leg extension.
  1 minute between each machine is planned.
  Other Names: 3/7 method
Other: Cardiac rehabilitation with 3X9 method — HIIT ( 2 min 80% wmax: 2 min 50% wmax) during 30 minutes 3X9 method 9 rep 1 minute of rest, 9 rep (1 min) and 9 rep (total volume : 27 repetitions) at 70 of 1 repetition Leg press, Dips Press, Leg curl, Traction and Leg extension.
  1 minute between each machine is planned
  Other Names: 3X9 method

SUMMARY:
The study proposes to measure the effect of resitance training (RT) (3/7 method) on biological markers of muscle hypertrophy in a cardiac population.

3/7 method consisting of five sets of an increasing number of repetitions (3 to 7) during successive sets and brief inter-set intervals (15 s). This method is compare to 3X9 method, 3 series of 9 repetitions with inter-set (1min).The training exercise consisted of contraction on machine (leg press, triceps press, leg curl, traction, leg extension) with load of ~ 70% of one repetition maximal (1RM).

Before these trainings all subject perform HIIT on bicycles (2 min high intensity (80% Wmax) and 2 min low intensity (50% Wmax) during 30 minutes.

The investigators collect blood sample before exercice, after HIIT and after RT.

It is randomized cross-over study.

DETAILED DESCRIPTION:
The subjects come on two different days minimum 2 days and maximum 10 days between the two tests. They were instructed to avoid exercise the day before they participated in the study.

The investigators collect blood 2 minutes after endurance training (HIIT) and 2 min after RT training.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Coronary artery diseases
* Heart failure with reduced ejection fraction

Exclusion Criteria:

* angina
* acutely decompensated heart failure
* electrocardiographic evidence of ischemia
* significant valvular disease
* orthopedic/neurologic disorders that limited exercise

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Change in Lactate | within 2 minutes after TR training session on day 1
  mmol/l
change in Testosterone | within 2 minutes after TR training session on day 1
  nmol/l
change Glucocorticoid Cortisol | within 2 minutes after TR training session on day 1
  nmol/l
change in Growth Hormone | within 2 minutes after TR training session on day 1
  ng/ml
change in ph | within 2 minutes after TR training session on day 1
  venoust
change PCO2 venoust | within 2 minutes after TR training session on day 1
  mm Hg

SECONDARY OUTCOMES:
Borg scale | within 4 minutes after TR training session on day 1
  Borg Rating of Perceived Exertion - Borg modified (0 = no exertion at all -10 maximal exertion)
Pleasure of the session scale | within 4 minutes after TR training session on day 1
  0 = worse 10 = better

CONTACTS AND LOCATIONS:
Overall Officials: Philippe van de borne, Professor, Study Director — Erasme University Hospital, Université Libre de Bruxelles, Brussels, Belgium
Locations (1):
- Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
on request

REFERENCES:
- [Background] Mang ZA, Realzola RA, Ducharme J, Bellissimo GF, Beam JR, Mermier C, de Castro Magalhaes F, Kravitz L, Amorim FT. The effect of repetition tempo on cardiovascular and metabolic stress when time under tension is matched during lower body exercise. Eur J Appl Physiol. 2022 Jun;122(6):1485-1495. doi: 10.1007/s00421-022-04941-3. Epub 2022 Apr 8. PMID 35394146